CLINICAL TRIAL: NCT01687218
Title: A Phase 2 Randomized Sequence Open Label Expanded Safety and Acceptability Study of Oral Emtricitabine/Tenofovir Disoproxil Fumarate Tablet and Rectally-Applied Tenofovir Reduced-Glycerin 1% Gel
Brief Title: Safety and Acceptability Study of Oral Emtricitabine/Tenofovir Disoproxil Fumarate Tablet and Rectally-Applied Tenofovir Reduced-Glycerin 1% Gel
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: CONRAD (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); National Institute of Mental Health (NIMH) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: MTN-017; 5UM1AI068633 (NIH); 11857 (Other: DAIDS protocol #)
Record Dates: First submitted 2012-08-27; First posted 2012-09-18 (Estimated); Results first posted 2017-02-01 (Estimated); Last update posted 2021-06-24 (Actual); Status verified 2021-06

CONDITIONS: HIV
MeSH Terms: interventions — Tenofovir; Gels

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Group 1 (Active Comparator): Daily Oral Emtricitabine/Tenofovir Disoproxil Fumarate Tablet (8 weeks); followed by Daily Rectally-Applied Tenofovir Reduced Glycerin 1% Gel (8 weeks); followed by Receptive Anal Intercourse Associated Rectally-Applied Tenofovir Reduced Glycerin 1% Gel (8 weeks)
  Interventions: Drug: Oral FTC/TDF (Daily Emtricitabine/Tenofovir Disoproxil fumarate Tablet); Drug: Rectal Daily TFV RG 1% gel (Rectally applied Tenofovir Reduced Glycerin 1% Gel); Drug: Rectal RAI-associated TFV RG 1% gel (Receptive Anal Intercourse Associated rectally applied Tenofovir Reduced Glycerin 1% Gel)
- Group 2 (Active Comparator): Receptive Anal Intercourse Associated Rectally-Applied Tenofovir Reduced Glycerin 1% Gel (8 weeks); followed by Daily Oral Emtricitabine/Tenofovir Disoproxil Fumarate Tablet (8 weeks); followed by Daily Rectally-Applied Tenofovir Reduced Glycerin 1% Gel (8 weeks)
  Interventions: Drug: Oral FTC/TDF (Daily Emtricitabine/Tenofovir Disoproxil fumarate Tablet); Drug: Rectal Daily TFV RG 1% gel (Rectally applied Tenofovir Reduced Glycerin 1% Gel); Drug: Rectal RAI-associated TFV RG 1% gel (Receptive Anal Intercourse Associated rectally applied Tenofovir Reduced Glycerin 1% Gel)
- Group 3 (Active Comparator): Daily Rectally-Applied Tenofovir Reduced Glycerin 1% Gel (8 weeks); followed by Receptive Anal Intercourse Associated Rectally-Applied Tenofovir Reduced Glycerin 1% Gel (8 weeks); followed by Daily Oral Emtricitabine/Tenofovir Disoproxil Fumarate Tablet (8 weeks)
  Interventions: Drug: Oral FTC/TDF (Daily Emtricitabine/Tenofovir Disoproxil fumarate Tablet); Drug: Rectal Daily TFV RG 1% gel (Rectally applied Tenofovir Reduced Glycerin 1% Gel); Drug: Rectal RAI-associated TFV RG 1% gel (Receptive Anal Intercourse Associated rectally applied Tenofovir Reduced Glycerin 1% Gel)
- Group 4 (Active Comparator): Daily Rectally-Applied Tenofovir Reduced Glycerin 1% Gel (8 weeks); followed by Daily Oral Emtricitabine/Tenofovir Disoproxil Fumarate Tablet (8 weeks); followed by Receptive Anal Intercourse Associated Rectally-Applied Tenofovir Reduced Glycerin 1% Gel (8 weeks)
  Interventions: Drug: Oral FTC/TDF (Daily Emtricitabine/Tenofovir Disoproxil fumarate Tablet); Drug: Rectal Daily TFV RG 1% gel (Rectally applied Tenofovir Reduced Glycerin 1% Gel); Drug: Rectal RAI-associated TFV RG 1% gel (Receptive Anal Intercourse Associated rectally applied Tenofovir Reduced Glycerin 1% Gel)
- Group 5 (Active Comparator): Daily Oral Emtricitabine/Tenofovir Disoproxil Fumarate Tablet (8 weeks); followed by Receptive Anal Intercourse Associated Rectally-Applied Tenofovir Reduced Glycerin 1% Gel (8 weeks); followed by Daily Rectally-Applied Tenofovir Reduced Glycerin 1% Gel (8 weeks)
  Interventions: Drug: Oral FTC/TDF (Daily Emtricitabine/Tenofovir Disoproxil fumarate Tablet); Drug: Rectal Daily TFV RG 1% gel (Rectally applied Tenofovir Reduced Glycerin 1% Gel); Drug: Rectal RAI-associated TFV RG 1% gel (Receptive Anal Intercourse Associated rectally applied Tenofovir Reduced Glycerin 1% Gel)
- Group 6 (Active Comparator): Receptive Anal Intercourse Associated Rectally-Applied Tenofovir Reduced Glycerin 1% Gel (8 weeks);followed by Daily Rectally-Applied Tenofovir Reduced Glycerin 1% Gel (8 weeks); followed by Daily Oral Emtricitabine/Tenofovir Disoproxil Fumarate Tablet (8 weeks)
  Interventions: Drug: Oral FTC/TDF (Daily Emtricitabine/Tenofovir Disoproxil fumarate Tablet); Drug: Rectal Daily TFV RG 1% gel (Rectally applied Tenofovir Reduced Glycerin 1% Gel); Drug: Rectal RAI-associated TFV RG 1% gel (Receptive Anal Intercourse Associated rectally applied Tenofovir Reduced Glycerin 1% Gel)

INTERVENTIONS:
Drug: Oral FTC/TDF (Daily Emtricitabine/Tenofovir Disoproxil fumarate Tablet)
Drug: Rectal Daily TFV RG 1% gel (Rectally applied Tenofovir Reduced Glycerin 1% Gel)
Drug: Rectal RAI-associated TFV RG 1% gel (Receptive Anal Intercourse Associated rectally applied Tenofovir Reduced Glycerin 1% Gel)

SUMMARY:
MTN-017 is a Phase 2, multi-site, randomized, six-sequence, two three-period, open label crossover study, examining the effects of oral Truvada and reduced glycerin 1% tenofovir gel. The study population will be sexually active, HIV-uninfected males who are 18 years of age or older, who report a history of receptive anal intercourse in the past 3 months. Each of the study product regimens offers different advantages to participants seeking an effective HIV prevention agent. How these relative advantages will compare in terms of safety, acceptability, systemic and local absorption, and adherence will be examined within this study.

ELIGIBILITY:
Inclusion Criteria:

1. Male or transgender female > age of 18 at Screening
2. Able and willing to provide written informed consent
3. HIV-1 uninfected at Screening and Enrollment
4. Able and willing to provide adequate locator information, as defined in site SOP
5. Available to return for all study visits, barring unforeseen circumstances and willing to comply with study participation requirements
6. In general good health at Screening and Enrollment, as determined by the site IoR or designee
7. Per participant report, a history of consensual RAI at least once in the past 3 months
8. Per participant report at Screening and Enrollment, agrees not to engage in receptive or insertive sexual activity with another study participant for the duration of study participation.
9. Willing to use study-provided condoms for the duration of the study for penetrative intercourse
10. Willing to not take part in other research studies involving drugs, medical devices, vaccines or genital products for the duration of study participation (including the time between Screening and Enrollment)
11. Men and transgender females who agree to take part in the PK, PD and Mucosal Immunology Subset, must also agree to abstain from:

    * Inserting anything into the rectum, including abstaining from RAI for 72 hours after the collection of biopsies
    * Taking non-steroidal anti-inflammatory drugs (NSAIDs), aspirin and/or other drugs that are associated with increased likelihood of bleeding following mucosal biopsy collection for 72 hours prior to and following the collection of biopsies.

Exclusion Criteria:

1. At Screening, participant-reported symptoms, and/or clinical or laboratory diagnosis of active anorectal or reproductive tract infection requiring treatment per current World Health Organization (WHO) guidelines or symptomatic urinary tract infection (UTI). Infections requiring treatment include symptomatic Chlamydia trachomatis (CT) infection, Neisseria gonorrhea (GC), syphilis, active herpes simplex virus (HSV) lesions, anogenital sores or ulcers, or symptomatic genital warts.

   Note: HSV-1 or HSV-2 seropositive diagnosis with no active lesions is allowed, since treatment is not required.

   In cases of non-anorectal GC/CT identified at screening, one re-screening 2 months after the screening visit will be allowed
2. History of inflammatory bowel disease as reported by participant history
3. At Screening:

   * Positive for hepatitis B surface antigen
   * Positive for hepatitis C antibody
   * Hemoglobin < 10.0 g/dL
   * Platelet count less than 100,000/mm3
   * White blood cell count < 2,000 cells/mm3 or > 15,000 cells/mm3
   * Calculated creatinine clearance less than 60 mL/min by the Cockcroft-Gault formula where creatinine clearance in mL/min = (140 - age in years) x (weight in kg) x (1 for male)/72 x (serum creatinine in mg/dL)
   * Serum creatinine > 1.3 x the site laboratory upper limit of normal (ULN)
   * Alanine transaminase (ALT) and/or aspartate aminotransferase (AST) > 2.5× the site laboratory ULN
   * PK, PD and Immunological Subset only: International normalized ratio (INR) > 1.5× the site laboratory ULN or partial thromboplastin time (PTT) > 1.25× the site laboratory ULN
4. Known allergy to methylparaben and/or propylparaben
5. Known allergy to any of the study products.
6. Per participant report, use of the following medications and/or products within 12 weeks prior to screening, and/or anticipated use or unwillingness to abstain from use throughout study participation:

   * Any investigational products
   * Systemic immunomodulatory medications
   * Use of Heparin, including Lovenox®
   * Warfarin
   * Plavix® (clopidogrel bisulfate)
   * Rectally-administered medications or products, containing N-9 or corticosteroids
7. By participant report, use of post-exposure prophylaxis (PEP) for HIV exposure within the 12 weeks prior to screening or anticipated use during study participation.
8. Symptoms suggestive of acute HIV seroconversion at Screening and Enrollment
9. Has any other condition that, in the opinion of the Investigator of Record (IoR)/designee, would preclude informed consent, make study participation unsafe, complicate interpretation of study outcome data, or otherwise interfere with achieving the study objectives would make the patient unsuitable for the study or unable/unwilling to comply with the study requirements. Such conditions may include, but are not limited to, colorectal abnormalities, substance abuse, or renal, hepatic, hematological, gastrointestinal, endocrine, pulmonary, neurological or psychiatric disease.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 195 (Actual)
Dates: Start 2013-09-25 (Actual); Primary Completion 2015-05-26 (Actual); Study Completion 2015-05-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ross D. Cranston, MD, FRCP, Study Chair — University of Pittsburgh Medical Center (UPMC); Javier R. Lama, MD, MPH, Study Chair — Asociacion Civil Impacta Salud y Educacion (IMPACTA)
Locations (8):
- United States (3):
  - HIV Research Section, San Francisco - Department of Public Health, San Francisco, California
  - The Fenway Institute/Fenway Community Health, Boston, Massachusetts
  - University of Pittsburgh Medical Center (UPMC), Pittsburgh, Pennsylvania
- Asociacion Civil Impacta Salud y Educacion (IMPACTA), Lima, Peru
- University of Puerto Rico Medical Sciences Campus - Maternal Infant Studies Center (CEMI), San Juan, Puerto Rico
- Desmond Tutu HIV Foundation, Cape Town, South Africa
- Thailand (2):
  - Research Institute for Health Sciences - Chiang Mai University, Chiang Mai
  - Thailand MOPH - US CDC Collaboration (TUC), Nonthaburi

REFERENCES:
- [Result] Cranston RD, Lama JR, Richardson BA, Carballo-Dieguez A, Kunjara Na Ayudhya RP, Liu K, Patterson KB, Leu CS, Galaska B, Jacobson CE, Parikh UM, Marzinke MA, Hendrix CW, Johnson S, Piper JM, Grossman C, Ho KS, Lucas J, Pickett J, Bekker LG, Chariyalertsak S, Chitwarakorn A, Gonzales P, Holtz TH, Liu AY, Mayer KH, Zorrilla C, Schwartz JL, Rooney J, McGowan I; MTN-017 Protocol Team. MTN-017: A Rectal Phase 2 Extended Safety and Acceptability Study of Tenofovir Reduced-Glycerin 1% Gel. Clin Infect Dis. 2017 Mar 1;64(5):614-620. doi: 10.1093/cid/ciw832. PMID 27986684
- [Result] Carballo-Dieguez A, Balan IC, Brown W 3rd, Giguere R, Dolezal C, Leu CS, Marzinke MA, Hendrix CW, Piper JM, Richardson BA, Grossman C, Johnson S, Gomez K, Horn S, Kunjara Na Ayudhya RP, Patterson K, Jacobson C, Bekker LG, Chariyalertsak S, Chitwarakorn A, Gonzales P, Holtz TH, Liu A, Mayer KH, Zorrilla C, Lama J, McGowan I, Cranston RD. High levels of adherence to a rectal microbicide gel and to oral Pre-Exposure Prophylaxis (PrEP) achieved in MTN-017 among men who have sex with men (MSM) and transgender women. PLoS One. 2017 Jul 27;12(7):e0181607. doi: 10.1371/journal.pone.0181607. eCollection 2017. PMID 28750059
- [Result] Giguere R, Brown W III, Balan IC, Dolezal C, Ho T, Sheinfil A, Ibitoye M, Lama JR, McGowan I, Cranston RD, Carballo-Dieguez A. Are participants concerned about privacy and security when using short message service to report product adherence in a rectal microbicide trial? J Am Med Inform Assoc. 2018 Apr 1;25(4):393-400. doi: 10.1093/jamia/ocx081. PMID 29025127
- [Result] Carballo-Dieguez A, Giguere R, Dolezal C, Leu CS, Balan IC, Brown W 3rd, Rael C, Richardson BA, Piper JM, Bekker LG, Chariyalertsak S, Chitwarakorn A, Gonzales P, Holtz TH, Liu A, Mayer KH, Zorrilla CD, Lama JR, McGowan I, Cranston RD; MTN-017 Protocol Team. Preference of Oral Tenofovir Disoproxil Fumarate/Emtricitabine Versus Rectal Tenofovir Reduced-Glycerin 1% Gel Regimens for HIV Prevention Among Cisgender Men and Transgender Women Who Engage in Receptive Anal Intercourse with Men. AIDS Behav. 2017 Dec;21(12):3336-3345. doi: 10.1007/s10461-017-1969-1. PMID 29119473
- [Result] Giguere R, Rael CT, Sheinfil A, Balan IC, Brown W 3rd, Ho T, Dolezal C, Leu CS, Liu A, Mayer KH, Lama JR, McGowan I, Carballo-Dieguez A, Cranston RD; MTN-017 Protocol Team. Factors Supporting and Hindering Adherence to Rectal Microbicide Gel Use with Receptive Anal Intercourse in a Phase 2 Trial. AIDS Behav. 2018 Feb;22(2):388-401. doi: 10.1007/s10461-017-1890-7. PMID 28825142
- [Result] Brown W 3rd, Giguere R, Sheinfil A, Ibitoye M, Balan I, Ho T, Brown B, Quispe L, Sukwicha W, Lama JR, Carballo-Dieguez A, Cranston RD. Challenges and solutions implementing an SMS text message-based survey CASI and adherence reminders in an international biomedical HIV PrEP study (MTN 017). J Biomed Inform. 2018 Apr;80:78-86. doi: 10.1016/j.jbi.2018.02.018. Epub 2018 Mar 6. PMID 29501908
- [Result] Cranston RD, Carballo-Dieguez A, Gundacker H, Richardson BA, Giguere R, Dolezal C, Siegel A, KunjaraNaAyudhya RP, Gomez K, Piper JM, Lama JR, McGowan I; MTN-017 Protocol Team. Prevalence and determinants of anal human papillomavirus infection in men who have sex with men and transgender women. Int J STD AIDS. 2019 Feb;30(2):154-162. doi: 10.1177/0956462418797864. Epub 2018 Oct 18. PMID 30336747
- [Result] Leu CS, Giguere R, Bauermeister JA, Dolezal C, Brown W 3rd, Balan IC, Richardson BA, Piper JM, Lama JR, Cranston RD, Carballo-Dieguez A. Trajectory of use over time of an oral tablet and a rectal gel for HIV prevention among transgender women and men who have sex with men. AIDS Care. 2019 Mar;31(3):379-387. doi: 10.1080/09540121.2018.1533223. Epub 2018 Oct 14. PMID 30318905
- [Result] Liu AY, Norwood A, Gundacker H, Carballo-Dieguez A, Johnson S, Patterson K, Bekker LG, Chariyalertsak S, Chitwarakorn A, Gonzales P, Holtz TH, Mayer KH, Zorrilla C, Buchbinder S, Piper JM, Lama JR, Cranston RD. Brief Report: Routine Use of Oral PrEP in a Phase 2 Rectal Microbicide Study of Tenofovir Reduced-Glycerin 1% Gel (MTN-017). J Acquir Immune Defic Syndr. 2019 Aug 15;81(5):516-520. doi: 10.1097/QAI.0000000000002066. PMID 31299013
- [Result] Balan IC, Giguere R, Brown W 3rd, Carballo-Dieguez A, Horn S, Hendrix CW, Marzinke MA, Ayudhya RPKN, Patterson K, Piper JM, McGowan I, Lama JR, Cranston RD; MTN-017 Protocol Team. Brief Participant-Centered Convergence Interviews Integrate Self-Reports, Product Returns, and Pharmacokinetic Results to Improve Adherence Measurement in MTN-017. AIDS Behav. 2018 Mar;22(3):986-995. doi: 10.1007/s10461-017-1955-7. PMID 29076032
- [Derived] McGowan IM, Kunjara Na Ayudhya RP, Brand RM, Marzinke MA, Hendrix CW, Johnson S, Piper J, Holtz TH, Curlin ME, Chitwarakorn A, Raengsakulrach B, Doncel G, Schwartz JL, Rooney JF, Cranston RD. An Open-Label Pharmacokinetic and Pharmacodynamic Assessment of Tenofovir Gel and Oral Emtricitabine/Tenofovir Disoproxil Fumarate. AIDS Res Hum Retroviruses. 2022 Apr;38(4):279-287. doi: 10.1089/AID.2021.0115. Epub 2021 Oct 29. PMID 34541872

RESULTS

PARTICIPANT FLOW:
Recruitment Details: HIV-uninfected males or transgender females who were 18 years of age or older who practice receptive anal intercourse were recruited from September 2013 through November 2014 from 8 sites in Peru, Puerto Rico, South Africa, Thailand and USA.
Pre-assignment Details: 349 persons were screened and 154 were excluded for various reasons. The study enrolled 195 participants, 187 of whom are evaluable. Evaluable participants are those participants who were enrolled and not replaced, or were the final enrolled replacement participant for another enrolled participant who met the criteria for replacement.
Groups:
- Group 1: Daily Oral Emtricitabine/Tenofovir Disoproxil Fumarate Tablet (8 weeks); followed by Daily Rectally-Applied Tenofovir Reduced Glycerin 1% Gel (8 weeks); followed by Receptive Anal Intercourse Associated Rectally-Applied Tenofovir Reduced Glycerin 1% Gel (8 weeks)
  Oral FTC/TDF (Daily Emtricitabine/Tenofovir Disoproxil fumarate Tablet)
  Rectal Daily TFV RG 1% gel (Rectally applied Tenofovir Reduced Glycerin 1% Gel)
  Rectal RAI-associated TFV RG 1% gel (Receptive Anal Intercourse Associated rectally applied Tenofovir Reduced Glycerin 1% Gel)
- Group 2: Receptive Anal Intercourse Associated Rectally-Applied Tenofovir Reduced Glycerin 1% Gel (8 weeks); followed by Daily Oral Emtricitabine/Tenofovir Disoproxil Fumarate Tablet (8 weeks); followed by Daily Rectally-Applied Tenofovir Reduced Glycerin 1% Gel (8 weeks)
  Oral FTC/TDF (Daily Emtricitabine/Tenofovir Disoproxil fumarate Tablet)
  Rectal Daily TFV RG 1% gel (Rectally applied Tenofovir Reduced Glycerin 1% Gel)
  Rectal RAI-associated TFV RG 1% gel (Receptive Anal Intercourse Associated rectally applied Tenofovir Reduced Glycerin 1% Gel)
- Group 3: Daily Rectally-Applied Tenofovir Reduced Glycerin 1% Gel (8 weeks); followed by Receptive Anal Intercourse Associated Rectally-Applied Tenofovir Reduced Glycerin 1% Gel (8 weeks); followed by Daily Oral Emtricitabine/Tenofovir Disoproxil Fumarate Tablet (8 weeks)
  Oral FTC/TDF (Daily Emtricitabine/Tenofovir Disoproxil fumarate Tablet)
  Rectal Daily TFV RG 1% gel (Rectally applied Tenofovir Reduced Glycerin 1% Gel)
  Rectal RAI-associated TFV RG 1% gel (Receptive Anal Intercourse Associated rectally applied Tenofovir Reduced Glycerin 1% Gel)
- Group 4: Daily Rectally-Applied Tenofovir Reduced Glycerin 1% Gel (8 weeks); followed by Daily Oral Emtricitabine/Tenofovir Disoproxil Fumarate Tablet (8 weeks); followed by Receptive Anal Intercourse Associated Rectally-Applied Tenofovir Reduced Glycerin 1% Gel (8 weeks)
  Oral FTC/TDF (Daily Emtricitabine/Tenofovir Disoproxil fumarate Tablet)
  Rectal Daily TFV RG 1% gel (Rectally applied Tenofovir Reduced Glycerin 1% Gel)
  Rectal RAI-associated TFV RG 1% gel (Receptive Anal Intercourse Associated rectally applied Tenofovir Reduced Glycerin 1% Gel)
- Group 5: Daily Oral Emtricitabine/Tenofovir Disoproxil Fumarate Tablet (8 weeks); followed by Receptive Anal Intercourse Associated Rectally-Applied Tenofovir Reduced Glycerin 1% Gel (8 weeks); followed by Daily Rectally-Applied Tenofovir Reduced Glycerin 1% Gel (8 weeks)
  Oral FTC/TDF (Daily Emtricitabine/Tenofovir Disoproxil fumarate Tablet)
  Rectal Daily TFV RG 1% gel (Rectally applied Tenofovir Reduced Glycerin 1% Gel)
  Rectal RAI-associated TFV RG 1% gel (Receptive Anal Intercourse Associated rectally applied Tenofovir Reduced Glycerin 1% Gel)
- Group 6: Receptive Anal Intercourse Associated Rectally-Applied Tenofovir Reduced Glycerin 1% Gel (8 weeks);followed by Daily Rectally-Applied Tenofovir Reduced Glycerin 1% Gel (8 weeks); followed by Daily Oral Emtricitabine/Tenofovir Disoproxil Fumarate Tablet (8 weeks)
  Oral FTC/TDF (Daily Emtricitabine/Tenofovir Disoproxil fumarate Tablet)
  Rectal Daily TFV RG 1% gel (Rectally applied Tenofovir Reduced Glycerin 1% Gel)
  Rectal RAI-associated TFV RG 1% gel (Receptive Anal Intercourse Associated rectally applied Tenofovir Reduced Glycerin 1% Gel)
Period: Overall Study
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Group 5 | Group 6
Started | 33 | 32 | 31 | 34 | 33 | 32
Completed | 30 | 29 | 30 | 32 | 32 | 32
Not Completed | 3 | 3 | 1 | 2 | 1 | 0
Not completed — Withdrawal by Subject | 2 | 3 | 0 | 1 | 1 | 0
Not completed — Relocated, no follow-up planned | 1 | 0 | 1 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Includes all participants enrolled.
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Group 5 | Group 6 | Total
Number analyzed (Participants) | 33 | 32 | 31 | 34 | 33 | 32 | 195
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.9 (8.5) | 30.4 (10.6) | 32.4 (9.2) | 29.6 (8.9) | 32.2 (10.6) | 31.4 (7.8) | 31.1 (9.3)
Age, Customized [Number; unit: participants]
  Under 20 | 2 | 1 | 2 | 1 | 2 | 2 | 10
  20-24 | 7 | 7 | 6 | 12 | 7 | 5 | 44
  25-29 | 7 | 11 | 6 | 6 | 7 | 6 | 43
  30-34 | 6 | 4 | 6 | 7 | 7 | 10 | 40
  35-39 | 6 | 4 | 2 | 2 | 2 | 4 | 20
  40-44 | 4 | 3 | 4 | 3 | 3 | 2 | 19
  45-49 | 0 | 0 | 4 | 2 | 2 | 3 | 11
  50+ | 1 | 2 | 1 | 1 | 3 | 0 | 8
Sex/Gender, Customized [Number; unit: participants] — One participant from Peru did not complete a baseline CASI.
  participants
    Man | 21 | 21 | 22 | 27 | 26 | 24 | 141
    Woman | 0 | 0 | 1 | 1 | 1 | 1 | 4
    Transgender/Transwoman | 4 | 6 | 2 | 3 | 3 | 1 | 19
    Other | 5 | 4 | 6 | 3 | 3 | 6 | 27
    Refuse to answer | 2 | 1 | 0 | 0 | 0 | 0 | 3
Hispanic Origin [Number; unit: participants]
  Yes | 10 | 9 | 8 | 8 | 12 | 8 | 55
  No | 23 | 23 | 23 | 26 | 21 | 24 | 140
Highest Level of Education [Number; unit: participants]
  no schooling | 0 | 0 | 0 | 0 | 0 | 0 | 0
  primary school, not complete | 0 | 0 | 0 | 1 | 0 | 0 | 1
  primary school, complete | 0 | 0 | 1 | 0 | 0 | 1 | 2
  secondary school, not complete | 2 | 1 | 1 | 1 | 3 | 1 | 9
  secondary school, complete | 2 | 5 | 6 | 4 | 4 | 6 | 27
  attended college or university | 29 | 26 | 23 | 28 | 26 | 24 | 156
Sexual Orientation (CASI) [Number; unit: participants] — One participant from Peru did not complete a baseline CASI.
  participants
    Gay/Homosexual | 27 | 26 | 27 | 32 | 28 | 31 | 171
    Bisexual | 3 | 3 | 3 | 0 | 3 | 1 | 13
    Straight/Heterosexual | 0 | 1 | 1 | 1 | 0 | 0 | 3
    Other | 1 | 1 | 0 | 1 | 2 | 0 | 5
    Refuse to answer | 1 | 1 | 0 | 0 | 0 | 0 | 2
Nationality [Number; unit: participants] — Country in which the site clinic resides.
  participants
    Puerto Rico | 1 | 1 | 1 | 1 | 2 | 1 | 7
    Peru | 7 | 6 | 6 | 6 | 7 | 6 | 38
    South Africa | 3 | 3 | 3 | 3 | 3 | 3 | 18
    Thailand | 9 | 9 | 9 | 9 | 9 | 9 | 54
    U.S.A. | 13 | 13 | 12 | 15 | 12 | 13 | 78
Race - Puerto Rico [Number; unit: participants]
  White | 0 | 0 | 0 | 0 | 2 | 0 | 2
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Mixed | 0 | 1 | 0 | 0 | 0 | 1 | 2
  Black | 0 | 0 | 1 | 1 | 0 | 0 | 2
  Indigenous | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Other | 1 | 0 | 0 | 0 | 0 | 0 | 1
Race - Peru [Number; unit: participants]
  White | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Mixed | 6 | 3 | 3 | 4 | 3 | 5 | 24
  Black | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Indigenous | 1 | 3 | 3 | 1 | 4 | 1 | 13
  Other | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race - South Africa [Number; unit: participants]
  Other African tribe | 0 | 0 | 0 | 1 | 0 | 1 | 2
  White | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Zulu | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Xhosa | 3 | 2 | 3 | 2 | 3 | 1 | 14
  Indian | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Colored | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Other | 0 | 1 | 0 | 0 | 0 | 0 | 1
Race - Thailand [Number; unit: participants]
  Indian | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Mixed | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Thai | 9 | 9 | 9 | 9 | 9 | 9 | 54
  Chinese | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Other | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race - U.S.A. [Number; unit: participants]
  White | 12 | 11 | 10 | 12 | 6 | 10 | 61
  Asian | 0 | 0 | 0 | 0 | 2 | 2 | 4
  Mixed | 0 | 0 | 0 | 0 | 2 | 0 | 2
  Black/African-American | 0 | 0 | 0 | 3 | 0 | 0 | 3
  American Indian/Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native-Hawaiian or other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Other | 1 | 2 | 2 | 0 | 2 | 1 | 8

OUTCOME MEASURES:

1. Primary Outcome: Safety: Grade 2 or Higher Adverse Events
Description: Compare the safety profiles of daily FTC/TDF tablet, daily TFV RG 1% gel, and RAI-associated TFV RG 1% gel. Analysis of the primary endpoint of grade 2 or higher AEs was performed on only the evaluable participants based on the principle of intent-to-treat (ITT) whereby participants who were randomized were included in the analysis regardless of whether or not they received product in a given period (i.e, were lost to follow-up, or terminated early and/or were on a product hold).
Time Frame: 27 weeks (three 8-week product use periods with 1-week washout periods between them)
Population: Among the 187 evaluable participants. One participant was terminated before the Initiate Period visit of his/her Period 3 (Oral Tablet regimen period). Thus, this participant is removed from the analysis of the oral period regimen.
Measure: Number; unit: participants
Groups:
- Product 1: Oral (Daily FTC/TDF)
- Product 2: Rectal (Daily TFV RG 1% gel)
- Product 3: Rectal (RAI-associated TFV RG 1% gel)
Arm/Group | Product 1 | Product 2 | Product 3
Number analyzed (Participants) | 186 | 187 | 187
participants | 64 | 61 | 56
Statistical Analysis 1: Comparison: Product 1 vs Product 2; Since some participants have more than one safety event per period of treatment regimen, a Generalized Estimating Equation (GEE) model with a Poisson (log) link, exchangeable correlation structure, and robust standard errors were used; Test type: Superiority or Other; p = 0.88, Generalized Estimating Equation (GEE); Risk Ratio (RR) = 1.03, 95% CI 2-sided [0.73 to 1.44] — It shows the rate ratio (RR) based on a GEE model comparing the Daily Rectal regimen with the Oral regimen and controlling for period in the model
Statistical Analysis 2: Comparison: Product 1 vs Product 3; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.43, Generalized Estimating Equation (GEE); Risk Ratio (RR) = 0.88, 95% CI 2-sided [0.64 to 1.21] — It shows the rate ratio (RR) based on a GEE model comparing the RAI Rectal regimen with the Oral regimen and controlling for period in the model

2. Primary Outcome: Acceptability: Participant Self-report of Liking the Product. H1-Overall How do You Feel About the Product You Used Recently?
Description: To evaluate and compare acceptability of daily FTC/TDF tablet, daily TFV RG 1% gel, and RAI-associated TFV RG 1% gel. Consistent with the acceptability endpoint of liking the product, a variable was created by combining from Section H. Liking the Product of the MTN-017 Follow-up Behavioral Questionnaire question 1A and question 1BC. Categories 1 and 2 were combined and categories 3 and 4 were combined to create a dichotomous variable.
Time Frame: 27 weeks (three 8-week product use periods with 1-week washout periods between them)
Population: All primary analyses are based on the data from evaluable participants. Evaluable participants are those participants who were enrolled and not replaced, or were the final enrolled replacement participant for another enrolled participant who met the criteria for replacement.
Measure: Number; unit: participants
Arm/Group | Product 1 | Product 2 | Product 3
Number analyzed (Participants) | 179 | 181 | 183
participants
  Disliked Very Much/A Little | 16 | 47 | 38
  Liked Very Much/A Little | 163 | 134 | 145
Statistical Analysis 1: Comparison: Product 1 vs Product 2; Generalized Estimating Equation (GEE) models with a binomial (logit) link, an exchangeable correlation structure and robust errors and with treatment regimen and period as independent variables were used to compare the three treatment regimens for the acceptability endpoints. The oral arm and period 1 were used as the reference group in each of the models; Test type: Superiority or Other; p < 0.0001, Generalized Estimating Equation (GEE); Odds Ratio (OR) = 0.28, 95% CI 2-sided [0.15 to 0.50] — Oral regimen is the reference group
Statistical Analysis 2: Comparison: Product 1 vs Product 3; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.002, Generalized Estimating Equation (GEE); Odds Ratio (OR) = 0.37, 95% CI 2-sided [0.20 to 0.70] — Oral regimen is the reference group

3. Primary Outcome: Acceptability: Participant Self-report of Ease of Use. I1-Overall How Easy or Difficult Was it to Use the Product?
Description: To evaluate and compare acceptability of daily FTC/TDF tablet, daily TFV RG 1% gel, and RAI-associated TFV RG 1% gel. Consistent with the acceptability endpoint of ease of use, a variable was created to compare regimens. This variable combines questions 1A and 1BC from Section I. Ease of Use of the MTN-017 Follow-up Behavioral Questionnaire. Categories 1 and 2 were combined and categories 3 and 4 were combined to create dichotomous variables.
Time Frame: 27 weeks (three 8-week product use periods with 1-week washout periods between them)
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Product 1 | Product 2 | Product 3
Number analyzed (Participants) | 183 | 184 | 183
participants
  Very Difficult/Difficult | 14 | 24 | 18
  Very Easy/Easy | 169 | 160 | 165
Statistical Analysis 1: Comparison: Product 1 vs Product 2; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.08, Generalized Estimating Equation (GEE); Odds Ratio (OR) = 0.56, 95% CI 2-sided [0.29 to 1.08] — Oral regimen is the reference group
Statistical Analysis 2: Comparison: Product 1 vs Product 3; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.46, Generalized Estimating Equation (GEE); Odds Ratio (OR) = 0.76, 95% CI 2-sided [0.37 to 1.56] — Oral regimen is the reference group

4. Primary Outcome: Acceptability: Participant Self-report of Likelihood of Product Use if Shown to be Effective. N1-If This Product Provides Some Protection How Likely Would You be to Take it?
Description: To evaluate and compare acceptability of daily FTC/TDF tablet, daily TFV RG 1% gel, and RAI-associated TFV RG 1% gel. Consistent with the acceptability endpoint of likelihood to use product in the future, a variable was created by combining Section N. Likelihood to Use Product in the Future of the MTN-017 Follow-up Behavioral Questionnaire questions 1A, 1B, and 1C. Categories 1 and 2 were combined and categories 3 and 4 were combined to create a dichotomous variable.
Time Frame: 27 weeks (three 8-week product use periods with 1-week washout periods between them)
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Product 1 | Product 2 | Product 3
Number analyzed (Participants) | 183 | 184 | 176
participants
  Very Unlikely/Unlikely | 24 | 52 | 31
  Very Likely/Likely | 159 | 132 | 145
Statistical Analysis 1: Comparison: Product 1 vs Product 2; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.0004, Generalized Estimating Equation (GEE); Odds Ratio (OR) = 0.38, 95% CI 2-sided [0.22 to 0.65] — Oral regimen is the reference group
Statistical Analysis 2: Comparison: Product 1 vs Product 3; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.23, Generalized Estimating Equation (GEE); Odds Ratio (OR) = 0.70, 95% CI 2-sided [0.39 to 1.25] — Oral regimen is the reference group

5. Secondary Outcome: Pharmacokinetics: Tenofovir (TFV) Concentrations (log10 ng/mL) in Blood Plasma
Description: Compare tenofovir concentrations in blood plasma among daily FTC/TDF tablet, daily TFV RG 1% gel, and RAI-associated TFV RG 1% gel groups.
Time Frame: 27 weeks (three 8-week product use periods with 1-week washout periods between them)
Population: Participant periods with tenofovir concentrations (log10 ng/mL) in blood plasma among evaluable participants.
Measure: Mean (Standard Deviation); unit: log10 ng/mL
Arm/Group | Product 1 | Product 2 | Product 3
Number analyzed (Participants) | 184 | 184 | 183
log10 ng/mL
  Mid-Period TFV Concentration: number analyzed (Participants) | 183 | 182 | 182
  Mid-Period TFV Concentration | 1.85 (0.59) | 0.42 (0.83) | -0.01 (0.89)
  End Period TFV Concentration: number analyzed (Participants) | 183 | 179 | 179
  End Period TFV Concentration | 1.77 (0.71) | 0.37 (0.84) | -0.02 (0.92)
Statistical Analysis 1: Comparison: Product 1 vs Product 2; Mixed effects models were used to compare the three treatment regimens within participants over time using the oral regimen as the reference group. The models included fixed effects for treatment regimen and period and random effects for participant within sequence. The log 10 transformation was used in the mixed effects models for all PK results to achieve normality; Test type: Other; p < 0.001, Mixed Models Analysis; Slope = -1.41, 95% CI 2-sided [-1.53 to -1.30] — This comparison is between the daily rectal and oral (reference) groups for tenofovir levels in blood plasma, log10 ng/mL
Statistical Analysis 2: Comparison: Product 1 vs Product 3; [analysis description as in outcome 5, analysis 1]; Test type: Other; p < 0.001, Mixed Models Analysis; Slope = -1.82, 95% CI 2-sided [-1.95 to -1.70] — This comparison is between the RAI rectal and oral (reference) groups for tenofovir levels in blood plasma, log10 ng/mL

6. Secondary Outcome: Pharmacokinetics: End Period Tenofovir (TFV) Concentrations (log10 ng/mg) in Rectal Tissue
Description: Compare end period tenofovir concentrations in rectal tissue among daily FTC/TDF tablet, daily TFV RG 1% gel, and RAI-associated TFV RG 1% gel groups.
Time Frame: 27 weeks (three 8-week product use periods with 1-week washout periods between them)
Population: Participant end periods with tenofovir concentrations (log10 ng/mg) in rectal tissue among evaluable participants.
Measure: Mean (Standard Deviation); unit: log10 ng/mg
Arm/Group | Product 1 | Product 2 | Product 3
Number analyzed (Participants) | 36 | 36 | 36
log10 ng/mg | 0.18 (0.51) | 0.84 (0.50) | 0.02 (0.87)
Statistical Analysis 1: Comparison: Product 1 vs Product 2; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p < 0.001, Mixed Models Analysis; Slope = 0.66, 95% CI 2-sided [0.49 to 0.83] — Oral regimen is the reference group
Statistical Analysis 2: Comparison: Product 1 vs Product 3; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p = 0.31, Mixed Models Analysis; Slope = -0.16, 95% CI 2-sided [-0.46 to 0.15] — Oral regimen is the reference group

7. Secondary Outcome: Pharmacokinetics: Tenofovir (TFV) Concentrations (log10 ng/mg) in Rectal Sponge
Description: Compare tenofovir concentrations in rectal sponge specimens among daily FTC/TDF tablet, daily TFV RG 1% gel, and RAI-associated TFV RG 1% gel groups.
Time Frame: 27 weeks (three 8-week product use periods with 1-week washout periods between them)
Population: Participant periods with tenofovir concentrations (log10 ng/mg) in rectal sponge specimens among evaluable participants.
Measure: Mean (Standard Deviation); unit: log10 ng/mg
Arm/Group | Product 1 | Product 2 | Product 3
Number analyzed (Participants) | 186 | 183 | 184
log10 ng/mg
  Initiate Period TFV Concentration: number analyzed (Participants) | 122 | 121 | 121
  Initiate Period TFV Concentration | -1.53 (1.20) | -1.65 (1.12) | -1.29 (1.42)
  Mid-Period TFV Concentration: number analyzed (Participants) | 183 | 180 | 183
  Mid-Period TFV Concentration | 0.71 (1.22) | 0.97 (1.64) | -0.03 (1.54)
  End Period TFV Concentration: number analyzed (Participants) | 183 | 175 | 178
  End Period TFV Concentration | 0.66 (1.31) | 1.00 (1.42) | 0.01 (1.67)
Statistical Analysis 1: Comparison: Product 1 vs Product 2; Mixed effects models were used to compare the three treatment regimens within participants over time using the oral regimen as the reference group. The models included fixed effects for treatment regimen and period and random effects for participant within sequence. The log 10 transformation was used in the mixed effects models for all PK results to achieve normality. Mid period and end period visits only were used in this analysis; Test type: Superiority; p = 0.004, Mixed Models Analysis; Slope = 0.30, 95% CI 2-sided [0.10 to 0.50]
Statistical Analysis 2: Comparison: Product 1 vs Product 3; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p < 0.001, Mixed Models Analysis; Slope = -0.70, 95% CI 2-sided [-0.92 to -0.47]

8. Secondary Outcome: Pharmacokinetics: Emtricitabine (FTC) Concentrations (log10 ng/mL) in Blood Plasma
Description: Compare emtricitabine concentrations in blood plasma among daily FTC/TDF tablet, daily TFV RG 1% gel, and RAI-associated TFV RG 1% gel groups.
Time Frame: 27 weeks (three 8-week product use periods with 1-week washout periods between them)
Population: Participant periods with emtricitabine (FTC) concentrations (log10 ng/mL) in blood plasma among evaluable participants.
Measure: Mean (Standard Deviation); unit: log10 ng/mL
Arm/Group | Product 1 | Product 2 | Product 3
Number analyzed (Participants) | 184 | 184 | 183
log10 ng/mL
  Mid-Period FTC Concentration: number analyzed (Participants) | 183 | 182 | 182
  Mid-Period FTC Concentration | 2.34 (0.82) | -0.35 (1.00) | -0.37 (0.98)
  End Period FTC Concentration: number analyzed (Participants) | 183 | 179 | 179
  End Period FTC Concentration | 2.25 (0.96) | -0.37 (0.98) | -0.33 (1.06)
Statistical Analysis 1: Comparison: Product 1 vs Product 2; Mixed effects models were used to compare the three treatment regimens within participants over time using the oral regimen as the reference group. The models included fixed effects for treatment regimen and period and random effects for participant within sequence. The log 10 transformation was used in the mixed effects models for all PK results to achieve normality for the following analysis; Test type: Superiority; p < 0.001, Mixed Models Analysis; Slope = -2.66, 95% CI 2-sided [-2.82 to -2.50]
Statistical Analysis 2: Comparison: Product 1 vs Product 3; [analysis description as in outcome 8, analysis 1]; Test type: Superiority; p < 0.001, Mixed Models Analysis; Slope = -2.65, 95% CI 2-sided [-2.81 to -2.49]

9. Secondary Outcome: Pharmacokinetics: End Period Emtricitabine (FTC) Concentrations (log10 ng/mg) in Rectal Tissue
Description: Compare end period emtricitabine concentrations in rectal tissue among daily FTC/TDF tablet, daily TFV RG 1% gel, and RAI-associated TFV RG 1% gel groups.
Time Frame: 27 weeks (three 8-week product use periods with 1-week washout periods between them)
Population: Participant end periods with emtricitabine (FTC) concentrations (log10 ng/mg) in rectal tissue among evaluable participants.
Measure: Mean (Standard Deviation); unit: log10 ng/mg
Arm/Group | Product 1 | Product 2 | Product 3
Number analyzed (Participants) | 36 | 36 | 36
log10 ng/mg | -0.35 (0.33) | -1.26 (0.00) | -1.26 (0.00)
Statistical Analysis 1: Comparison: Product 1 vs Product 2; Mixed effects models were used to compare the three treatment regimens within participants over time using the oral regimen as the reference group. The models included fixed effects for treatment regimen and period and random effects for participant within sequence. The log 10 transformation was used in the mixed effects models for all PK results to achieve normality. End period visits only are used in this analysis; Test type: Superiority; p < 0.001, Mixed Models Analysis; Slope = -0.91, 95% CI 2-sided [-1.01 to -0.80]
Statistical Analysis 2: Comparison: Product 1 vs Product 3; [analysis description as in outcome 9, analysis 1]; Test type: Superiority; p < 0.001, Mixed Models Analysis; Slope = -0.91, 95% CI 2-sided [-1.01 to -0.80]

10. Secondary Outcome: Pharmacokinetics: Emtricitabine (FTC) Concentrations (log10 ng/mg) in Rectal Sponge
Description: Compare emtricitabine concentrations in rectal sponge among daily FTC/TDF tablet, daily TFV RG 1% gel, and RAI-associated TFV RG 1% gel groups.
Time Frame: 27 weeks (three 8-week product use periods with 1-week washout periods between them)
Population: Participant periods with emtricitabine (FTC) concentrations (log10 ng/mg) in rectal sponge specimens among evaluable participants.
Measure: Mean (Standard Deviation); unit: log10 ng/mg
Arm/Group | Product 1 | Product 2 | Product 3
Number analyzed (Participants) | 186 | 183 | 184
log10 ng/mg
  Initiate Period FTC Concentration: number analyzed (Participants) | 121 | 122 | 120
  Initiate Period FTC Concentration | -1.75 (0.80) | -1.76 (0.73) | -1.57 (1.00)
  Mid-Period FTC Concentration: number analyzed (Participants) | 183 | 180 | 182
  Mid-Period FTC Concentration | 0.31 (1.14) | -1.76 (0.76) | -1.67 (0.91)
  End Period FTC Concentration: number analyzed (Participants) | 183 | 175 | 178
  End Period FTC Concentration | 0.14 (1.30) | -1.80 (0.69) | -1.69 (0.87)
Statistical Analysis 1: Comparison: Product 1 vs Product 2; Mixed effects models were used to compare the three treatment regimens within participants over time using the oral regimen as the reference group. The models included fixed effects for treatment regimen and period and random effects for participant within sequence. The log 10 transformation was used in the mixed effects models for all PK results to achieve normality. Mid period and end period visits only are used in this analysis; Test type: Superiority; p < 0.001, Mixed Models Analysis; Slope = -2.00, 95% CI 2-sided [-2.16 to -1.84]
Statistical Analysis 2: Comparison: Product 1 vs Product 3; [analysis description as in outcome 10, analysis 1]; Test type: Superiority; p < 0.001, Mixed Models Analysis; Slope = -1.90, 95% CI 2-sided [-2.07 to -1.74]

11. Secondary Outcome: Pharmacokinetics: End Period Tenofovir-Diphosphate (TFV-DP) Concentrations (log10 ng/mg) in Rectal Tissue
Description: Compare end period tenofovir-diphosphate (TFV-DP) concentrations in rectal tissue among daily FTC/TDF tablet, daily TFV RG 1% gel, and RAI-associated TFV RG 1% gel groups.
Time Frame: 27 weeks (three 8-week product use periods with 1-week washout periods between them)
Population: Participant end periods with tenofovir-diphosphate (TFV-DP) concentrations (log10 ng/mg) in rectal tissue among evaluable participants.
Measure: Mean (Standard Deviation); unit: log10 ng/mg
Arm/Group | Product 1 | Product 2 | Product 3
Number analyzed (Participants) | 36 | 36 | 36
log10 ng/mg | 1.52 (0.50) | 2.06 (0.52) | 1.54 (0.92)
Statistical Analysis 1: Comparison: Product 1 vs Product 2; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p < 0.001, Mixed Models Analysis; Slope = 0.54, 95% CI 2-sided [0.35 to 0.72]
Statistical Analysis 2: Comparison: Product 1 vs Product 3; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p = 0.92, Mixed Models Analysis; Slope = 0.01, 95% CI 2-sided [-0.28 to 0.31]

12. Secondary Outcome: Adherence: Percentage of Prescribed Doses Taken Orally or Administered Rectally in an 8-week Period
Description: Compare percentage of prescribed doses taken orally or administered rectally in an 8-week period based on the Final Converged Rates. Final Converged Rates were measured first via self-report through Short Message Service (SMS). The clinic staff also reported the most likely number of doses taken. Finally, the MTN Behavioral Research Working Group (BRWG) provided the final estimate of the number of doses taken for each participant for each period based on self-report, staff estimates and PK testing results. Note that these final judgement data are missing if PK results are missing.
Time Frame: 27 weeks (three 8-week product use periods with 1-week washout periods between them)
Population: Evaluable participants with Final Converged Rates of prescribed doses.
Measure: Count of Participants; unit: Participants
Arm/Group | Product 1 | Product 2 | Product 3
Number analyzed (Participants) | 185 | 184 | 183
Participants
  Less Than 80% | 12 | 31 | 13
  At or Greater than 80% | 173 | 153 | 170
Statistical Analysis 1: Comparison: Product 1 vs Product 2; Generalized Estimating Equation (GEE) models with a binomial (logit) link, an exchangeable correlation structure and robust errors and with treatment regimen and period as independent variables was used to compare the three treatment regimens for the acceptability endpoints. Because the distribution of the adherence percentages were skewed, we did not use a linear mixed effects model as originally planned. Instead, we dichotomized the adherence percentage into<80% adherence versus>80% adherence; Test type: Superiority; p = 0.0005, Generalized Estimating Equations (GEE); Odds Ratio (OR) = 0.35, 95% CI 2-sided [0.19 to 0.63] — Oral regimen is the reference group
Statistical Analysis 2: Comparison: Product 1 vs Product 3; [analysis description as in outcome 12, analysis 1]; Test type: Superiority; p = 0.74, Generalized Estimating Equations (GEE); Odds Ratio (OR) = 0.89, 95% CI 2-sided [0.43 to 1.81] — Oral regimen is the reference group

13. Other Pre Specified Outcome: Pharmacodynamics
Description: To characterize pharmacodynamic responses following oral and rectal exposure to antiretroviral drugs
Time Frame: 27 weeks (three 8-week product use periods with 1-week washout periods between them)
Reporting Status: Not Posted

14. Other Pre Specified Outcome: Mucosal Immunity
Description: To characterize changes in mucosal immunity between baseline and the end of the daily FTC/TDF and TFV RG 1% gel product use
Time Frame: 27 weeks (three 8-week product use periods with 1-week washout periods between them)
Reporting Status: Not Posted

15. Other Pre Specified Outcome: Correlation Between PK and Adherence
Description: To assess correlation of PK with adherence measures
Time Frame: 27 weeks (three 8-week product use periods with 1-week washout periods between them)
Reporting Status: Not Posted

16. Other Pre Specified Outcome: Factors Associated With Adherence
Description: To identify factors associated with product adherence and whether they differ by product used (FTC/TDF or TFV RG 1% gel) or regimen (daily use or RAI-associated use)
Time Frame: 27 weeks (three 8-week product use periods with 1-week washout periods between them)
Reporting Status: Not Posted

17. Other Pre Specified Outcome: Sexual Activity and Condom Use
Description: To examine whether sexual activity or condom use varies by product used
Time Frame: 27 weeks (three 8-week product use periods with 1-week washout periods between them)
Reporting Status: Not Posted

18. Other Pre Specified Outcome: Product Sharing
Description: To determine the level of sharing of study products with non-participants and to assess with whom products are shared
Time Frame: 27 weeks (three 8-week product use periods with 1-week washout periods between them)
Reporting Status: Not Posted

19. Other Pre Specified Outcome: Problem Practices
Description: To determine the prevalence of behavioral practices associated with anal intercourse that may affect microbicide use
Time Frame: 27 weeks (three 8-week product use periods with 1-week washout periods between them)
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 27 weeks (three 8-week product use periods with 1-week washout periods between them)
Description: AEs are reported throughout follow-up. AEs are assigned to a regimen based on the reported or derived onset date being on or after the first visit of the regimen and before the start of the next regimen.
Arm/Group | Product 1 | Product 2 | Product 3
Serious Adverse Events (participants affected / at risk) | 1/192 | 2/192 | 0/191
Other Adverse Events (participants affected / at risk) | 85/192 | 103/192 | 87/191
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Product 1 (N=192) | Product 2 (N=192) | Product 3 (N=191)
Hospitalisation (Surgical and medical procedures) | 0 | 1 | 0
Appendicitis (Infections and infestations) | 0 | 1 | 0
Suicide attempt (Psychiatric disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Product 1 (N=192) | Product 2 (N=192) | Product 3 (N=191)
Abdominal distension (Gastrointestinal disorders) | 4 | 2 | 6
Abdominal pain (Gastrointestinal disorders) | 8 | 5 | 7
Anal fissure (Gastrointestinal disorders) | 1 | 7 | 7
Anorectal discomfort (Gastrointestinal disorders) | 0 | 6 | 3
Defaecation urgency (Gastrointestinal disorders) | 2 | 16 | 11
Diarrhoea (Gastrointestinal disorders) | 14 | 22 | 15
Dyspepsia (Gastrointestinal disorders) | 7 | 3 | 0
Flatulence (Gastrointestinal disorders) | 12 | 23 | 14
Gastrointestinal mucosa hyperaemia (Gastrointestinal disorders) | 1 | 6 | 2
Nausea (Gastrointestinal disorders) | 15 | 4 | 2
Proctalgia (Gastrointestinal disorders) | 3 | 7 | 4
Rectal haemorrhage (Gastrointestinal disorders) | 4 | 9 | 5
Rectal tenesmus (Gastrointestinal disorders) | 0 | 7 | 3
Vomiting (Gastrointestinal disorders) | 6 | 4 | 1
Fatigue (General disorders) | 6 | 1 | 2
Nasopharyngitis (Infections and infestations) | 12 | 10 | 20
Proctitis chlamydial (Infections and infestations) | 9 | 8 | 13
Proctitis gonococcal (Infections and infestations) | 5 | 3 | 6
Upper respiratory tract infection (Infections and infestations) | 5 | 10 | 11
Viral upper respiratory tract infection (Infections and infestations) | 7 | 11 | 10
Dizziness (Nervous system disorders) | 9 | 3 | 6
Headache (Nervous system disorders) | 17 | 9 | 7
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 6 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No